CLINICAL TRIAL: NCT03818763
Title: Phase I Study Evaluating Safety and Feasibility of Hematopoietic Stem Cell Gene Transfer That Targets Factor VIII Delivery From Platelets for Patients With Hemophilia A
Brief Title: Gene Therapy Trial for Platelet Derived Factor VIII Production in Hemophilia A
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Mary Eapen MBBS MS, Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00033763
Record Dates: First submitted 2019-01-15; First posted 2019-01-28 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Hemophilia A
Keywords: Gene Therapy
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Intervention Model Description: Open-label, nonrandomized, single-center phase I cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous CD34+PBSC transduced with a lentiviral vector (Experimental): Patients will receive a patient specific (autologous) cytokine mobilized CD34+Peripheral Blood Stem Cells (PBSC) transduced ex vivo with a lentiviral vector containing cDNA encoding the human B-domain deleted FVIII protein.
  Interventions: Biological: Auto CD34+PBSC, transduced with a lentiviral vector encoding the B domain deleted from of human coagulation factor VIII

INTERVENTIONS:
Biological: Auto CD34+PBSC, transduced with a lentiviral vector encoding the B domain deleted from of human coagulation factor VIII — Reduced intensity conditioning with melphalan and fludarabine, followed by a single infusion of autologous CD34+PBSC, transduced with a lentiviral vector (-889ITGA2B-BDDFVIII-WPTS(MUT6)(VSVg)) also known as (Pleightlet(MUT6)) encoding the B domain deleted from of human coagulation factor VIII (BDDFVIII) in up to five hemophilia A patients with a history of FVIII inhibitors (≥0.6BU).
  The infusion volume of transduced cells will not exceed 20 ml/kg body weight.

SUMMARY:
This is a Phase I study. This research study is being conducted to find new ways to treat severe hemophilia A. This study is a gene therapy study. Gene therapy is an experimental way to introduce, into a person's cells, specific genetic material. A gene can be delivered/introduced into a cell using a carrier known as a "vector." In this study, a virus (lentivirus), the "vector", is used to introduce or deliver a gene that creates and stores a protein Factor VIII (FVIII) in your platelets. These platelets are made from stem cells (mother cells for your bone marrow) that are removed from your blood by a procedure called apheresis. This research study will take some of the patient's own stem cells, from the apheresis procedure, and genetically modify them using the vector in order to make them produce FVIII in platelets that arise from the stem cells. They will then give the genetically modified stem cells back to the patient so that they can possibly create platelets that produce and store Factor VIII on their own.

DETAILED DESCRIPTION:
This is an open label, nonrandomized, single center, phase I cohort study, involving reduced intensity conditioning, followed by a single infusion of autologous CD34+PBSC, transduced with a lentiviral vector (-889ITGA2B-BDDFVIII-WPTS (MUT6)(VSVg)) also known as (Pleightlet(MUT6)) encoding the B domain deleted from of human coagulation factor VIII (BDDFVIII) in up to five hemophilia A patients with a history of FVIII inhibitors (≥0.6BU) .

ELIGIBILITY:
Inclusion Criteria:

Study population will include: adult males >18 years of age with a diagnosis of severe hemophilia A and currently active or a history of FVIII inhibitors (≥0.6 BU). Females will be excluded because hemophilia A is an X-linked disorder that is extremely rare in females.

1. Confirmed diagnosis of severe hemophilia A by undetectable plasma factor VIII:C by a one-stage PTT-based assay and coatest chromogenic factor VIII assay. Subjects with currently active or a history of positive FVIII inhibitor titers (≥0.6 BU) irrespective of their titer or current inhibitor status will be included for enrollment.
2. Subject may be prescribed prophylactic therapy with factor VIII bypassing agents or factor VIII mimetics prior to referral for inclusion in the study.
3. Subjects who are treated on demand using factor VIII bypassing agents must have a history of four or more bleeding episodes requiring treatment in the six-month period prior to referral for inclusion in the study.
4. Adequate bone marrow reserve as demonstrated by ANC >1.5/cu.mm; Hemoglobin >9g/dL; Platelets >100,000/microliter.
5. Adequate renal function, defined as creatinine clearance>60 ml/min (Cockroft-Gault formula)
6. Adequate liver function, defined as defined as total bilirubin ≤1.5 times the upper limit of normal (ULN) (excluding Gilbert's syndrome), both AST and ALT ≤3 times ULN at the time of screening, and no clinical signs or known laboratory/radiographic evidence consistent with cirrhosis.
7. Subject must sign an informed consent after explanation of the study and having questions answered.
8. Subject must be willing and able to document type of bleeding episodes and treatment in a paper or electronic diary during the study.
9. Subject must be willing to return for regular follow-up visits during the 15-year study.

Exclusion Criteria:

* A potential subject who meets any of the following exclusion criteria is ineligible to participate in the study.

  1. Therapy with factor VIII with the intent of immune tolerance induction within 30 days prior to inclusion within the study.
  2. Enrollment in another interventional clinical trial within 60 days prior to study inclusion.
  3. Medical contraindication to PBSC cytokine mobilization, use of GCSF, PBSC apheresis procedure or conditioning regimen.
  4. Medically significant organ dysfunction that would prevent compliance with conditioning or would severely limit the probability of survival based on clinical status.
  5. Those with a known co-existing clinically significant thrombophilic disorder, or as determined by the presence of any of the below identified on screening laboratory assessments:

     * FV Leiden
     * Protein S deficiency
     * Protein C deficiency
     * Prothrombin mutation (G20210A)
     * D-dimer >3 x the upper limit of normal (ULN) at Screening All known patients with the above and any patient with a personal or significant family history of thrombotic events (DVT, PE, arterial clots) as deemed by the principal investigator will be screened for the above disorders.
  6. Active invasive malignancy (Non-melanoma skin cancers and carcinoma in situ are not excluded).
  7. Known bone marrow disorders or abnormal bone marrow cytogenetics.
  8. Fertile males who are unwilling to use contraceptive techniques during and for the twelve months following treatment.
  9. Life expectancy severely limited by disease(s) other than hemophilia A.
  10. Patients with HIV, hepatitis B, hepatitis C (with an AST/ALT > 3 times the upper limit of normal).
  11. Other active infectious disease that is a contraindicat ion for immunosuppressive therapy.
  12. Patients who have elective surgery scheduled during the study period.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 5 (Estimated)
Dates: Start 2020-04-29 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2033-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of enrolled participants with adequate gene transduced hematopoietic stem cells for FVIII gene therapy infusion | Through study completion, an average of 4 years
  Assessed by availability of ≥4x106 transduced clinical grade CD34+PBSC per kg meeting release criteria for infusion; undetectable microbiological contamination and cell viability ≥70%.

SECONDARY OUTCOMES:
Incidence of toxicity from gene therapy | Within 3 months of gene therapy infusion
  Number of events meeting CTCAE criteria grade 3 or 4 toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Mary Eapen, MD, Principal Investigator — Froedtert Hosptial and Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States